CLINICAL TRIAL: NCT00973661
Title: Electronic Tools to Assist With Identification of and Counseling for Overweight Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Dr. Joyce Tang, Northwestern University, Department of General Internal Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00013264
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Overweight
Keywords: Overweight; Diagnosis; Counseling; Medical Records Systems, Computerized
MeSH Terms: conditions — Overweight; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic tools (Experimental)
  Interventions: Behavioral: Electronic tool set for counseling overweight patients
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Electronic tool set for counseling overweight patients — Physicians randomized to the "electronic tools" arm will receive access to a tool set to aid with counseling of overweight patients. This tool set includes the following components: automatic calculation of BMI, alert for overweight status, counseling template for weight loss goal-setting, linkage to referral options, and access to relevant patient handouts. Physicians randomized to the "usual care" arm will not receive access to these tools, and will continue to provide their usual care for overweight patients.
  Arms: Electronic tools

SUMMARY:
The purpose of this study is to design and assess the impact of an electronic alert and tool set to assist with physician identification and counseling of overweight patients.

DETAILED DESCRIPTION:
Overweight adults (Body Mass Index [BMI] 25-29.9) are at high risk for developing obesity, but rates of physician identification and counseling of overweight adults are low. Alerts and tools embedded in the electronic medical record have shown promise in enhancing quality improvement efforts.

Our aim is to design and assess the impact of an electronic alert and tool set to assist with identification and counseling of overweight patients with a BMI 27-29.9. Although the category of overweight patients spans BMI 25-29.9, we are including only patients with BMI 27-29.9 in order to focus resources on the most at-risk pre-obese population.

We will develop a tool set including the following components: automatic calculation of BMI, alert for overweight status, counseling template for weight loss goal-setting, linkage to referral options, and access to relevant patient handouts. Physicians in the Northwestern Memorial Faculty Foundation General Internal Medicine (NMFF GIM) practice who consent to participate in the study will be randomized into two groups, with one group of physicians receiving access to these tools. The other group of physicians will continue to provide their usual care for overweight patients. Outcome measures will include the following: tool usage; documentation of overweight in the problem list, encounter diagnosis, or note text; counseling for overweight and documentation of specific behavioral goals. Measures will be obtained via retrospective chart review.

ELIGIBILITY:
Inclusion Criteria (physicians):

* Consenting physicians from the Northwestern Memorial General Internal Medicine (NMFF GIM) practice

Exclusion Criteria (physicians):

* Study investigators will be excluded from participation (Dr. David Baker, Dr. Joyce Tang)

Inclusion Criteria (patients):

* Adults ages 18-65 seen at the NMFF GIM who are patients of consenting physicians
* Have at least one appointment at the NMFF GIM clinic between 9/1/09-2/28/10
* Body mass index (BMI) 27-29.9 at one or more visits between 9/1/09-2/28/10

Exclusion Criteria (patients):

* Patients without at least one recorded height measurement from any prior visit or without weight information from a visit within the 6 month target window will be excluded due to inability to calculate BMI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Documented diagnosis of overweight | September 1, 2009-February 28, 2010

SECONDARY OUTCOMES:
Documented counseling for overweight. | September 1, 2009-February 28, 2010
Documentation of specific behavior change goals | September 1, 2009-February 28, 2010

CONTACTS AND LOCATIONS:
Overall Officials: Joyce W Tang, MD, Principal Investigator — Northwestern University, Department of General Internal Medicine
Locations (1):
- Northwestern Memorial Faculty Foundation General Internal Medicine Clinic, Chicago, Illinois, United States